CLINICAL TRIAL: NCT02745392
Title: Randomized, Double-blind, Multi-center, Parallel-group, Dose-ranging Comparison of the Safety and Efficacy of the ZP-Zolmitriptan Intracutaneous Microneedle Systems to Placebo for the Acute Treatment of Migraine
Brief Title: Safety and Efficacy of ZP-Zolmitriptan Intracutaneous Microneedle Systems for the Acute Treatment of Migraine
Acronym: Zotrip
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-2016-001
Record Dates: First submitted 2016-04-14; First posted 2016-04-20 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Acute Migraine
Keywords: migraine; migraine headache; acute migraine; acute migraine headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ZP-Zolmitriptan 1 mg (Experimental): ZP-Zolmitriptan 1 mg patch single administration
  Interventions: Drug: ZP-Zolmitriptan
- ZP-Zolmitriptan 1.9 mg (Experimental): ZP-Zolmitriptan 1.9 mg patch single administration
  Interventions: Drug: ZP-Zolmitriptan
- ZP-Zolmitriptan 3.8 mg (Experimental): ZP-Zolmitriptan 3.8 mg (1.9 mg x 2 patches) single administration
  Interventions: Drug: ZP-Zolmitriptan
- Placebo (Placebo Comparator): Placebo (either single or double patch) single administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZP-Zolmitriptan — ZP-Zolmitriptan single administration delivered via intracutaneous microneedle patch delivery system
  Arms: ZP-Zolmitriptan 1 mg; ZP-Zolmitriptan 1.9 mg; ZP-Zolmitriptan 3.8 mg
Drug: Placebo — Placebo patch(es) to match ZP-Zolmitriptan single administration delivered via intracutaneous microneedle patch delivery system (one or two patches)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multi-center, parallel-group study designed to compare the safety and efficacy of a range of doses of ZP-Zolmitriptan intracutaneous microneedle systems to placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multi-center, parallel group study designed to compare the safety and efficacy of a range of doses of ZP-Zolmitriptan intracutaneous microneedle systems to placebo. Subjects who have consented and meet the entry criteria will be randomized to one of four blinded treatment groups. There will be a screening period of up to 1 week, followed by a run-in period to record migraine activity. The run-in period is to determine eligibility for randomization, and is planned to be 4 weeks in duration but may be extended up to an additional 4 weeks to accommodate scheduling. Qualified subjects will randomize to the double-blind treatment period at Day 0 and will have up to 8 weeks to confirm and treat a qualifying migraine. Using the eDiary to confirm they are experiencing a qualified migraine, subjects will self-administer the patch or patches and continue to respond to questions in the eDiary for 48 hours post treatment administration.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 1 year history of episodic, acute migraine (with or without aura) with onset prior to 50 years of age. Diagnosis must comply with International Headache Society (IHS) diagnostic criteria. Diagnostic criteria must include a history of at least five attacks not attributed to any other disorder that include all of the following criteria:

  1. Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
  2. Headache has at least two of the following characteristics:

  (i) unilateral location (ii) pulsating quality (iii) moderate or severe pain intensity (iv) aggravation by or causing avoidance of routine physical activity (e.g., walking or climbing stairs) c) During headache at least one of the following: (i) nausea and/or vomiting (ii) both photophobia and phonophobia
* Migraine history during the 6-month period prior to the run-in period must include: 2-8 migraines per month and no more than 10 headache days per month
* Women of child-bearing potential must not be pregnant, must agree to avoid pregnancy during the trial, and must use an acceptable methods of birth control for the duration of the trial.
* No significant ECG findings, defined by:

  1. ischemic changes
  2. Q-waves in at least two contiguous leads,
  3. clinically significant intra-ventricular conduction abnormalities (left bundle branch block or Wolf-Parkinson-White syndrome), or
  4. clinically significant arrhythmias (e.g., current atrial fibrillation)
* Able to understand the operation of the electronic diary and is able to apply the demo study drug patch.

Exclusion Criteria:

* Contraindication to triptans
* Use of any prohibited concomitant medications within 10 days of the Run-in Period
* History of hemiplegic or basilar migraine
* Participation in another investigational trial during the 30 days prior to the Run-in Period or during this study
* Previous participation in a clinical trial of ZP-Zolmitriptan
* Diagnosis of cancer (other than non-invasive skin cancer) within the 5 years prior to the Run-in Period
* History of unstable psychiatric illness requiring medication or hospitalization in the 12 months prior to the Run-in Period
* Subjects who have known allergy or sensitivity to zolmitriptan or its derivatives or formulations
* Subjects who have known allergy or sensitivity to adhesives
* Planned participation in activities which cause inflammation, irritation, sunburn, lesions, or tattoos at the intended application site from two weeks prior to screening through the last day of study participation
* Use of opiate analgesics or barbiturates more frequently than one day/week
* Women who are pregnant, breast-feeding or plan a pregnancy during this study
* Clinically significant liver disease
* Clinically significant kidney disease
* History of coronary artery disease (CAD), coronary vasospasm (including Prinzmetal's angina), aortic aneurysm, peripheral vascular disease or other ischemic diseases (e.g., ischemic bowel syndrome or Raynaud's syndrome)
* Three or more of the following CAD risk factors:

  * Current tobacco use
  * Hypertension or receiving anti-hypertensive medication for treatment of hypertension
  * Hyperlipidemia or on prescribed anti-cholesterol treatment
  * Family history of premature coronary artery disease (< 55 years of age in male first degree relatives or < 65 years of age in female first degree relatives)
  * Diabetes mellitus
* History of cerebral vascular accident, transient ischemic attacks, or seizures
* Hospitalization within the 30 days prior to the Run-in Period
* Any other household member currently participating in a ZP-Zolmitriptan study or relatives of site staff
* Any reason to believe that compliance with the study requirements and completion of evaluations required for this study will not be possible
* History or current abuse or dependence on alcohol or drugs that would interfere with adherence to study requirements
* Any clinically relevant abnormal findings in the physical exam, vital signs or laboratory tests that, in the opinion of the Investigator, may put the subject at risk

To be eligible for Treatment, subjects must continue to meet all eligibility criteria and the following criteria observed during the Run-in Period:

1. An average of at least two qualifying migraines per 28-day period
2. No more than 10 headache days in the last 28 days prior to randomization
3. Demonstrated ability to properly use the eDiary and apply the demo study drug patch
4. Confirmation of continuing good general health, or stable non-serious disease that in the opinion of the Investigator will not place the subject at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Kellerman, Pharm.D., Study Director — Zosano Pharma Corporation
Locations (36):
- United States (36):
  - Clinical Research Advantage, Inc./Thunderbird Internal Medicine, Glendale, Arizona
  - The Research Center of Southern California, Carlsbad, California
  - Allergy and Asthma Specialists Medical Group and Research Center, Huntington Beach, California
  - Downtown LA Research Center, Los Angeles, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Empire Clinical Research, Upland, California
  - Colorado Allergy & AsthmaCenters, PC, Denver, Colorado
  - Ki Health Partners, Stamford, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Meridien Research, Tampa, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Boston Clinical Trials, Boston, Massachusetts
  - Novex Medical Research, New Bedford, Massachusetts
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Michigan Head Pain &Neurological Institute, Ann Arbor, Michigan
  - Westside Family Medical Center, P.C, Kalamazoo, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Clinvest/A Division of Banyan Group Inc., Springfield, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Nebraska Medical Research Institute, Bellevue, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Headache Wellness Center, PC, Greensboro, North Carolina
  - Peters Medical Research LLC, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Nashville Neurosciences Group, Nashville, Tennessee
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Charlottesville Medical Research Center LLC, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tepper SJ, Dodick DW, Schmidt PC, Kellerman DJ. Efficacy of ADAM Zolmitriptan for the Acute Treatment of Difficult-to-Treat Migraine Headaches. Headache. 2019 Apr;59(4):509-517. doi: 10.1111/head.13482. Epub 2019 Jan 30. PMID 30698272
- [Derived] Spierings EL, Brandes JL, Kudrow DB, Weintraub J, Schmidt PC, Kellerman DJ, Tepper SJ. Randomized, double-blind, placebo-controlled, parallel-group, multi-center study of the safety and efficacy of ADAM zolmitriptan for the acute treatment of migraine. Cephalalgia. 2018 Feb;38(2):215-224. doi: 10.1177/0333102417737765. Epub 2017 Oct 12. PMID 29022755

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | ZP-Zolmitriptan 1 mg | ZP-Zolmitriptan 1.9 mg | ZP-Zolmitriptan 3.8 mg
Started | 91 | 90 | 92 | 92
Completed | 91 | 89 | 92 | 92
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: mITT population
Groups:
- Placebo: Either single or double patch administration
- ZP-Zolmitriptan 1 mg: Single 1 mg patch administration
- ZP-Zolmitriptan 1.9 mg: Single 1.9 mg patch administration
- ZP-Zolmitriptan 3.8 mg: Double 1.9 mg patch administration
- Total: Total of all reporting groups
Arm/Group | Placebo | ZP-Zolmitriptan 1 mg | ZP-Zolmitriptan 1.9 mg | ZP-Zolmitriptan 3.8 mg | Total
Number analyzed (Participants) | 77 | 79 | 83 | 82 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.53) | 41.7 (11.58) | 40.1 (10.92) | 41.0 (11.39) | 41.3 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 73 | 68 | 280
  Male | 8 | 9 | 10 | 14 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 14 | 15 | 53
  Not Hispanic or Latino | 66 | 66 | 69 | 67 | 268
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 1 | 3 | 4 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 15 | 16 | 20 | 10 | 61
  White | 59 | 58 | 54 | 67 | 238
  More than one race | 2 | 1 | 3 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Pain Freedom
Description: Pain Freedom at 2 hours post study drug administration is one of the co-primary endpoints. Subjects were queried via their eDiary about their level of migraine pain (none, mild, moderate, or severe) at various intervals post-dose. Subjects who answered none at 2 hours post study drug were considered pain free at 2 hours.
Time Frame: 2 hours
Population: mITT population includes all subjects who were randomized, received any amount of study drug (applied the patch(es) to treat a qualifying migraine, and had at least 1 post-treatment efficacy assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ZP-Zolmitriptan 1 mg | ZP-Zolmitriptan 1.9 mg | ZP-Zolmitriptan 3.8 mg
Number analyzed (Participants) | 77 | 79 | 83 | 82
Participants | 11 | 24 | 23 | 34

2. Primary Outcome: Proportion of Subjects With Freedom From Most Bothersome Pre-specified Other Symptom (Nausea, Photophobia, or Phonophobia Pre-specified by Subject)
Description: The proportion of subjects with freedom from the subject's pre-specified most bothersome symptom at 2 hours is one of two parts of the co-primary efficacy endpoint. This endpoint will be evaluated separately but both endpoints have to be met statistically for the study to be considered a success.
Time Frame: 2 hours
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ZP-Zolmitriptan 1 mg | ZP-Zolmitriptan 1.9 mg | ZP-Zolmitriptan 3.8 mg
Number analyzed (Participants) | 77 | 79 | 83 | 82
Participants | 33 | 45 | 44 | 56

ADVERSE EVENTS:
Time Frame: 2-8 days post-study drug administration for a single migraine
Description: The number of subjects at risk includes only subjects who treated with study drug (333). Although 365 subjects were randomized, not all subjects had a migraine (a criterion for administering study drug) between randomization and the end of the trial. 32 subjects (8 in the placebo group, 10 in ZP-Zolmitriptan 1 mg, 5 in ZP-Zolmitriptan 1.9 mg, 9 in ZP-Zolmitriptan 3.8 mg) did not treat with study drug, and that is the difference between the number of subjects randomized and the number at risk.
Arm/Group | Placebo | ZP-Zolmitriptan 1 mg | ZP-Zolmitriptan 1.9 mg | ZP-Zolmitriptan 3.8 mg
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/80 | 0/87 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/80 | 0/87 | 0/83
Other Adverse Events (participants affected / at risk) | 15/83 | 26/80 | 37/87 | 43/83
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | ZP-Zolmitriptan 1 mg (N=80) | ZP-Zolmitriptan 1.9 mg (N=87) | ZP-Zolmitriptan 3.8 mg (N=83)
Application site erythema (General disorders) | 12 | 23 | 31 | 38
Application site bruise (General disorders) | 3 | 5 | 12 | 12
Application site pain (General disorders) | 1 | 2 | 2 | 8
Application site haemorrhage (General disorders) | 0 | 3 | 5 | 4
Application site swelling (General disorders) | 3 | 1 | 3 | 2
Application site oedema (General disorders) | 0 | 1 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 4
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less